CLINICAL TRIAL: NCT05212870
Title: Investıgatıon Of The Effect Of The Pandemıc Process On Cognıtıve Level, Paın Catastrophızatıon, Physıcal Actıvıty Level And Qualıty Of Lıfe In Indıvıduals Wıth Chronıc Low Back And Neck Paın
Brief Title: Investıgatıon Of The Effect Of The Pandemıc Process In Indıvıduals Wıth Chronıc Low Back And Neck Paın
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Professor, Physiotherapist, Hacettepe University
Other Study IDs: 16969557-1040
Record Dates: First submitted 2021-10-08; First posted 2022-01-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-08

CONDITIONS: Neck Pain; Low Back Pain; Cognitive Level; COVID-19 Pandemic
MeSH Terms: conditions — Neck Pain; Low Back Pain; COVID-19 | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back and neck pain group with experience of Covid-19
  Interventions: Other: assessment of cognitive level, pain catastrophe, physical activity level and quality of life
- Low back and neck pain group without experience of Covid-19
  Interventions: Other: assessment of cognitive level, pain catastrophe, physical activity level and quality of life

INTERVENTIONS:
Other: assessment of cognitive level, pain catastrophe, physical activity level and quality of life — assessment of cognitive level, pain catastrophe, physical activity level and quality of life

SUMMARY:
There are a limited number of studies examining the difficulty of reaching treatment related to the pandemic process and the general effects of the process in patients with chronic low back and neck pain. However, no study has been found that compares the effects of individuals actively carrying and not carrying the Covid-19 virus. For this reason, the aim of the study is to examine the effects of the pandemic process on the cognitive level, pain catastrophization, physical activity level and quality of life in individuals with chronic low back and neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-60,
* Having low back or neck pain lasting longer than 3 months,
* Having a history of Covid-19 (At least 6 weeks-post acute),
* Individuals with chronic low back and neck pain without a history of Covid-19 will be included.

Exclusion Criteria:

* Those with an active diagnosis of Covid-19
* Having a rheumatological disease,
* Broken etc. severe deformity that may lead to nerve injury,
* Having a history of spinal surgery,
* Having neurological disease in addition to spinal pathology,
* Having problems such as cancer, diabetes, dementia, organic brain dysfunction,
* Illiterate individuals will not be included.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic low back and neck pain
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Severity Assessment- Visual Analog Sacle | through study completion, an average of 1 year
  VAS indicates the level of pain that the person is currently experiencing with a vertical line on a plane. The pain felt by the person is marked as "0: I do not feel any pain", "10: I feel very severe pain". Scoring is based on measuring the vertical marking of the participant for pain marked on the plane with a ruler. The validity and reliability study of the scale was done by Price et al. made by

SECONDARY OUTCOMES:
Assessment of Cognitive Level: Montreal Cognitive Assessment Scale (MOCA) | 5 minutes, through study completion, an average of 1 year
  The scale consists of 11 questions in total. The score range is 0-30. Below 21 points is interpreted as cognitive disability for the Turkish population. Turkish validity and reliability study was conducted by Selekler et al. made by
Evaluation of Pain Catastrophization Level: Pain Catastrophization Scale | 5 minutes, through study completion, an average of 1 year
  There are 13 questions in total on this scale. The questions are aimed at questioning the feelings and thoughts of individuals during pain. Each question scores between 0 and 4. A score of 30 and above indicates the presence of pain catastrophization. The validity and reliability study of the Turkish version of the scale was conducted by Süren et al. made by.
Assessment of Physical Activity Level: International Physical Activity Questionnaire (UFAA)-Short Form | 5 minutes, through study completion, an average of 1 year
  It was developed by Craig, Marshall, Sjostrom, Bauman, and Booth (2003) by conducting validity and reliability studies of individuals in 12 different countries. The questionnaire is a valid tool developed to determine the physical activity levels of individuals between the ages of 18-65. There are eight versions of the questionnaire, which was adapted into Turkish by Öztürk (2005). It has been developed as four short and four long forms. The short form "last 7 days" was used in this study. The short form (7 questions) provides information about time spent walking, moderate-to-vigorous and vigorous activities. The time spent sitting is considered as a separate question. It is classified as low, medium and high level by calculating the activity level of the person in terms of METs according to the duration, frequency and intensity level of the movement.
Quality of Life Assessment: SF-36 | 5 minutes, through study completion, an average of 1 year
  SF-36 is a 36-item scale that evaluates the health status of a person with 8 sub-items (physical function, role limitations, social function, mental health, vitality, pain, general health). Each sub-item is scored separately between 0-100. As the score approaches 100, it indicates good health. Turkish validity and reliability study, Koçyiğit et al. (1999).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)